CLINICAL TRIAL: NCT03115710
Title: The K-Map Study, Global Prevalence of KC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: ELZA Institute (Unknown)
Responsible Party: Principal Investigator, Farhad Hafezi, MDPhD, University Hospital, Geneva
Other Study IDs: CR-09
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Keratoconus
Keywords: Keratoconus; Prevalence
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Rotating Scheimpflug camera (Pentacam HR) — One visit to Ophthalmology Department is required from participant. Parents or legal guardians must attend with their child. The interview and test during visit take approximately 15 minutes. Interview includes filling out a questionnaire about risk factors of the disease and double check on understanding the consent form. The child will sit in front of the instrument (Pentacam HR Scheimpflug imaging system). The rotational measuring procedure generates Scheimpflug images in three dimensions. The images taken during the examination are digitalized, and all image data are transferred to the computer. It calculates a 3D virtual model of the anterior eye segment, from which all additional information is derived.

SUMMARY:
Keratoconus is a ocular disease classified under ectatic diseases which often results in bilateral and asymmetrical corneal distortion. It usually affects patients at young age and can cause severe visual loss.

The overall goal of this study is to assess the prevalence of keratoconus (KC) in children and adolescents in various regions of the world based on modern tomographic imaging methods, and to verify whether the occurrence rates reported from literature should be corrected. Our hypothesis is that the prevalence of the disease is much higher than that traditionally reported.

At each site, corneal tomography examinations (Pentacam) will be performed bilaterally in children and adolescents, who are not ill or with any ophthalmological symptom. The population to be studied will be composed of children and adolescents on medical visits for non-ophthalmologic reasons, aged between 6 and 20 years. Multiple cities, from different continents (North America, South America, Asia and Europe) will participate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6-23 years of age.
* Subjects seen for a non-ophthalmic appointment
* Provide signed and dated patient consent form (signed by parents / legal guardians).
* Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

* Patients with a preexisting ocular disease / condition
* Pregnancy or breastfeeding

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This project will include children and adolescent age (6 - 23).The rationale for selecting this age range is to detect the disease KC at early stages.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2015-12-28 (Actual); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of keratoconus | 15 minutes
  Number of keratoconus cases detected

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Hafezi, Study Director — ELZA Institute
Locations (12):
- USC Roski Eye Institute, Los Angeles, California, United States
- Eye Hospital of Wenzhou Medical College, Wenzhou, China
- Zagreb, Croatia
- Alexandria, Egypt
- Homburg, Germany
- Isfahan, Iran
- Amman, Jordan
- Monterrey, Mexico
- Lima, Peru
- Ufa Eye Research Intitute, Ufa, Russia
- King Saud University, Riyadh, Saudi Arabia
- Bukhara, Uzbekistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres Netto EA, Al-Otaibi WM, Hafezi NL, Kling S, Al-Farhan HM, Randleman JB, Hafezi F. Prevalence of keratoconus in paediatric patients in Riyadh, Saudi Arabia. Br J Ophthalmol. 2018 Oct;102(10):1436-1441. doi: 10.1136/bjophthalmol-2017-311391. Epub 2018 Jan 3. PMID 29298777